CLINICAL TRIAL: NCT01174784
Title: A Non-randomized Study of the Avinger Wildcat Used to Cross Femoropopliteal CTOs
Brief Title: Chronic Total Occlusion Crossing With the Wildcat Catheter
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avinger, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVI CTO 10001
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Results first posted 2013-09-27 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Chronic Total Occlusions; Superficial Femoral Artery; Popliteal Artery
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): The Wildcat catheter is a CTO crossing catheter. Subjects will be subjected to crossing with this device.
  Interventions: Device: Chronic TOtAl OcclusioN CrossiNg with thE WildCat CatheTer

INTERVENTIONS:
Device: Chronic TOtAl OcclusioN CrossiNg with thE WildCat CatheTer — A Non-Randomized Study of the Avinger Wildcat™ used to Cross Chronic Total Occlusions in the Superficial Femoral and Popliteal Arteries
  Other Names: CONNECT

SUMMARY:
This is a prospective, multi-center, non-randomized study of the Wildcat Catheter to cross a single femoropopliteal chronic total occlusion (CTO). Safety and efficacy will be evaluated during the index procedure through 30-day follow-up.

DETAILED DESCRIPTION:
Patients with a CTO, defined as 99% to 100% stenosis of a peripheral artery, will be approached for enrollment in the study. Following providing informed consent, the CTO will be addressed by the Wildcat catheter, which will provide a route for the advancement of guidewires and other tools beyond the CTO. Data will be collected to assess the safety efficacy of use of the device during the procedure and up to 30 days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing and able to provide informed consent.
2. Patient is willing and able to comply with the study protocol.
3. Patient is > 18 years old.
4. Patient has peripheral arterial disease requiring revascularization as evidenced by contrast, CT or MR angiography.
5. Patient has an occluded femoropopliteal artery that is 99-100% stenosed and is ≥ 1 cm and ≤ 30 cm in length by visual estimate.
6. Target femoropopliteal vessel is ≥ 3.0 mm in diameter.
7. Patient has Rutherford Classification of 2-5.

Exclusion Criteria:

1. Patient has a known sensitivity or allergy to contrast materials that cannot be adequately pre-treated.
2. Patient has a known sensitivity or allergy to anti-platelet medications.
3. Patient is pregnant or lactating.
4. Patient has a co-existing disease or medical condition contraindicating percutaneous intervention.
5. Target vessel is severely calcified as evidenced by angiography.
6. Target lesion is in a bypass graft.
7. Target lesion is in a stent (i.e., in-stent restenosis).
8. Patient has had a procedure on the target limb within 7 days.
9. Patient has had a procedure on the target limb within the past 30 days and is unstable.
10. Patient is simultaneously participating in an investigational device or drug study.
11. Patient has a planned surgical or interventional procedure within 30 days after the study procedure.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Davis, MD, Principal Investigator — St. John Hospital; Laiq Raja, MD, Principal Investigator — El Paso Cardiology Associates
Locations (15):
- United States (15):
  - Birmingham Heart Clinic, Birmingham, Alabama
  - Arizona Regional / Adventis, Mesa, Arizona
  - Phoenix Heart Center, Phoenix, Arizona
  - Sutter Memorial, Sacramento, California
  - Sharp Memorial, San Diego, California
  - Coastal Vascular, Pensacola, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Detroit Medical Center, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Central Michigan Community Hospital, Mount Pleasant, Michigan
  - St. Louis University, St Louis, Missouri
  - Jobst Vascular Center, Toledo, Ohio
  - Austin Heart, Austin, Texas
  - Cardiology Care Consultants, El Paso, Texas
  - El Paso Cardiology Associates, El Paso, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited/enrolled in the study starting on August 31, 2010. 88 subjects were enrolled and exited the study by April 11, 2011. Angiographic review after the case revealed that 4 of the 88 cases did not meet the inclusion criteria and were considered screen failures per the protocol and excluded from the efficacy analyses.
Groups:
- Device Treatment: This is a one-arm study. All subjects will have a CTO addressed by the Wildcat crossing device.
Period: Overall Study
Arm/Group | Device Treatment
Started | 88
Completed | 84 (While 88 subjects did complete the procedure, 4 were considered screen failures post-procedure.)
Not Completed | 4
Not completed — Screen fails | 4

BASELINE CHARACTERISTICS:
Groups:
- Enrolled/Primary Cohort: Subjects with a CTO upon presentation to the surgical unit.
Arm/Group | Enrolled/Primary Cohort
Number analyzed (Participants) | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 47
Region of Enrollment [Number; unit: participants]
  United States | 88

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Events
Description: The primary safety endpoint of the CONNECT Study was defined as absence of in-hospital or 30-days Major Adverse Events (MAEs), no evidence of clinically significant perforations, clinically significant embolizations or Grade C or greater dissections after Wildcat CTO crossing confirmed by angiography.
Time Frame: Index through 30-Day Follow-Up
Population: Patients treated with Wildcat post guidewire failure.
Measure: Number; unit: participants
Groups:
- Enrolled/Primary Cohort: Patients with 99% to 100% stenosis of a peripheral artery were approached to join the study.
Arm/Group | Enrolled/Primary Cohort
Number analyzed (Participants) | 84
participants | 4

2. Primary Outcome: CTO Crossing Success Using the Wildcat
Description: Successful femoropopliteal CTO crossing using the Wildcat identified by confirmation of guidewire placement in the distal true lumen confirmed by angiography.
Time Frame: Index through 30-Day Follow-Up
Population: Patients treated with Wildcat post guidewire failure.
Measure: Number; unit: participants
Groups:
- Enrolled/Primary Cohort: Single arm in which the device was used
Arm/Group | Enrolled/Primary Cohort
Number analyzed (Participants) | 84
participants | 75

ADVERSE EVENTS:
Time Frame: 30-Days
Groups:
- Enrolled/Primary Cohort: Patient with 99% to 100% stenosis of a peripheral artery.
Arm/Group | Enrolled/Primary Cohort
Serious Adverse Events (participants affected / at risk) | 4/84
Other Adverse Events (participants affected / at risk) | 0/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled/Primary Cohort (N=84)
Major Adverse Event - Death (General disorders) | 0 (0)
Major Adverse Event - Unplanned Major Amputation (Vascular disorders) | 0 (0)
Major Adverse Event - Emergent Target Vessel Revascularization (Vascular disorders) | 0 (0)
Clinically Significant Perforation (Vascular disorders) | 4 (4)
Clinically Significant Embolization (Vascular disorders) | 0 (0)
Grade C Dissection (Vascular disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less